CLINICAL TRIAL: NCT03369106
Title: Mechanisms of Disease Severity in Multiple Sclerosis: an Integrative Multimodal Study
Acronym: SEP-BIO-PROG
Status: Active, not recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C16-114; 2017-A01844-49 (Registry Identifier: RCB)
Record Dates: First submitted 2017-11-28; First posted 2017-12-11 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Multiple Sclerosis siblings: Group of siblings having multiple sclerosis, n=120 Composite severity score calculation for all subjects
  Interventions: Other: Composite severity score calculation

INTERVENTIONS:
Other: Composite severity score calculation — Neurological examination, cognitive testing, and MRI exam

SUMMARY:
This study will identify a combination of disease severity markers (genetic, immunology, epigenetic, imaging) associated with disease severity and progression in a cohort of patients with multiple sclerosis.

DETAILED DESCRIPTION:
The heterogeneity of multiple sclerosis evolution relies on several pathophysiological mechanisms including neuroinflammation, neurodegeneration and remyelination and repair mechanisms.

The study will identify markers of disease severity in a longitudinal cohort of patients with multiple sclerosis who are siblings (both siblings having multiple sclerosis) including: biological markers (genetic, immunological and epigenetic markers, advanced MRI markers). An integrative model to predict disease progression will be proposed based on multimodal markers.

ELIGIBILITY:
Inclusion Criteria:

* Clinically isolated syndrome or Multiple sclerosis (2010 Mc Donald criteria)
* Sibling having Clinically isolated syndrome or Multiple sclerosis (2010 Mc Donald criteria) willing to participate to the study
* Affiliated to the French social security or equivalent

Exclusion Criteria:

* Cyclophosphamide, mitoxantrone or methylprednisolone infusion within one month before inclusion
* Multiple sclerosis relapse within one month before inclusion
* Concomitant severe or uncontrolled disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple Sclerosis siblings Group of siblings having multiple sclerosis, n=120
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-02-06 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
Change of Expanded Disability Status Scale (EDSS) | Baseline and 18 months
  Change in the Expanded Disability Status Scale (EDSS) which is the neurological assessment of disability related to multiple sclerosis.
  The EDSS measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. Scoring is based on measures of impairment in eight functional systems on examination by a neurologist.

SECONDARY OUTCOMES:
Change in neuropsychological scores | Baseline and 18 months
  Change in the battery of neuropsychological tests adapted for multiple sclerosis
Change in T2 lesion volume | Baseline and 18 months
  Change in volume of T2 lesion in the white matter
Grey matter volume change | Baseline and 18 months
  Change in cerebral grey matter volume

CONTACTS AND LOCATIONS:
Overall Officials: Céline Louapre, MD, PhD, Principal Investigator — Institut du Cerveau et de la Moelle Epinière
Locations (1):
- CIC Neurosciences Institut du Cerveau et de la Moelle Epinière, Paris, France

IPD SHARING:
Plan to Share IPD: No